CLINICAL TRIAL: NCT07358455
Title: Identification of Pre-prosthetic Revision Markers Predictive of Outcome in Patients With Periprosthetic Infection
Brief Title: Preop Biomarkers as Outcome Predictors in 2 Stage Revision Surgery for PJI
Acronym: ARKO-PJI
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7818
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Periprosthetic Joint Infection (PJI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With the progressive ageing of the population, a significant increase in the incidence of skeletal fractures-particularly of the proximal femur-as well as degenerative conditions such as osteoarthritis has been observed, for which joint arthroplasty represents the treatment of choice. However, this procedure is not free from complications; beyond technical and mechanical issues related to potential implant malpositioning, one of the most feared is periprosthetic joint infection (PJI), which poses a major challenge in terms of clinical management and prognostic impact. Therapeutic strategies for PJI range from debridement with retention of the implant and exchange of modular components (DAIR/DAPRI) to complete implant removal with insertion of an articulating spacer, often followed by a subsequent reimplantation procedure. These approaches require prolonged antibiotic regimens, potentially exerting a negative effect on renal function, particularly in cases of extended exposure to nephrotoxic agents. Despite the clinical relevance of this issue, the current literature still provides limited evidence regarding the identification of inexpensive and readily available biomarkers capable of predicting treatment outcomes in PJI, especially in patients undergoing spacer implantation followed by reimplantation. Recent literature has increasingly explored the use of biomarkers such as the neutrophil-to-lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR), monocyte-to-lymphocyte ratio (MLR), systemic inflammation response index (SIRI), and others to characterize inflammatory and nutritional status, and to investigate possible associations between these markers and the outcomes of selected surgical procedures. The availability of predictive markers could optimize therapeutic management by reducing the risk of infection recurrence and improving postoperative risk stratification.

ELIGIBILITY:
Inclusion criteria

* Age ≥ 18 years
* Diagnosis of an orthopaedic periprosthetic joint infection (PJI)
* Surgical treatment
* Minimum follow-up of 12 months
* Written informed consent to participate in the study

Exclusion criteria

* Age < 18 years
* Patients undergoing prosthetic revision without evidence of periprosthetic joint infection
* Treatment with antibiotic therapy alone (non-surgical management)
* Follow-up < 12 months
* Incomplete dataset
* Lack of informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PJI
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Biomarkers' capacity to predict the likelihood of prosthetic reimplantation | From enrollment for at least one year
  The ability of selected preoperative biomarkers (e.g., NLR, PLR) to predict reimplantation outcomes in patients undergoing two-stage revision procedures

SECONDARY OUTCOMES:
Acute kidney injury | From enrollment for at least one year
  Incidence of acute kidney injury
ADL/IADL | From enrollment for at least one year
  Activities of Daily Living (ADL) assess basic self-care functions (e.g., bathing, dressing, feeding, toileting, transferring), whereas Instrumental Activities of Daily Living (IADL) evaluate more complex skills required for independent living (e.g., managing medications, finances, transportation, shopping, meal preparation)
SF-12 | From enrollment for at least one year
  The 12-Item Short Form Health Survey (SF-12) is a validated patient-reported outcome measure that provides a concise assessment of health-related quality of life, generating two summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS)

REFERENCES:
- [Background] Tarabichi S, Lizcano JD, Abe EA, Goh GS, Baker CM, Parvizi J. Finding the Optimal Screening Test for Periprosthetic Joint Infection: A Prospective Study. J Arthroplasty. 2024 Aug;39(8):1919-1925.e2. doi: 10.1016/j.arth.2024.02.030. Epub 2024 Mar 6. PMID 38452860
- [Background] Jones IA, Wier J, Chen MS, Liu KC, Palmer R, Mayfield CK, Heckmann ND. Complete Blood Count Ratios Predict Adverse Events After Total Joint Arthroplasty. J Am Acad Orthop Surg. 2024 Dec 15;32(24):e1315-e1323. doi: 10.5435/JAAOS-D-24-00184. Epub 2024 Jun 6. PMID 38861722
- [Background] Balato G, Ascione T, Festa E, Di Gennaro D, Pandolfo G, Pagliano P. The Diagnostic Accuracy of Neutrophils to Lymphocytes Ratio, Platelets to Lymphocytes Ratio, Monocytes to Lymphocytes Ratio, and Platelets to Mean Platelet Volume Ratio in Diagnosing Periprosthetic Knee Infections. Are Gender-Specific Cutoff Values Needed? J Arthroplasty. 2023 May;38(5):918-924. doi: 10.1016/j.arth.2022.11.014. Epub 2022 Dec 5. PMID 36481284
- [Background] Ascione T, Balato G, Pagliano P. Upcoming evidence in clinical practice of two-stage revision arthroplasty for prosthetic joint infection. J Orthop Traumatol. 2024 May 18;25(1):26. doi: 10.1186/s10195-024-00767-1. PMID 38761247
- [Background] Zhang QY, Li HX, Xie HQ, Liu LM, Chen L, Zeng Y. Identifying potential predictive indicators for reimplantation timing in two-stage revision: a meta-analysis and system review. Arch Orthop Trauma Surg. 2024 Dec 23;145(1):88. doi: 10.1007/s00402-024-05689-5. PMID 39714508
- [Background] Karlidag T, Zanna L, Mundhe A, Gehrke T, Citak M. Admission Lymphocyte-to-C-Reactive Protein Ratio Predicts 90-Day Adverse Outcomes Following Aseptic Revision Total Hip Arthroplasty. J Arthroplasty. 2025 Nov 7:S0883-5403(25)01430-5. doi: 10.1016/j.arth.2025.11.004. Online ahead of print. PMID 41207340
- [Background] Muscaritoli M, Molfino A, Orlando S, Tambaro F. Assessing systemic inflammation and its prognostic value: Glasgow Prognostic Score, neutrophil-to-lymphocyte ratio or other options? Curr Opin Clin Nutr Metab Care. 2025 Sep 1;28(5):367-372. doi: 10.1097/MCO.0000000000001151. Epub 2025 Aug 1. PMID 40772508
- [Background] Parvizi J, Tan TL, Goswami K, Higuera C, Della Valle C, Chen AF, Shohat N. The 2018 Definition of Periprosthetic Hip and Knee Infection: An Evidence-Based and Validated Criteria. J Arthroplasty. 2018 May;33(5):1309-1314.e2. doi: 10.1016/j.arth.2018.02.078. Epub 2018 Feb 26. PMID 29551303
- [Background] Mu W, Xu B, Wang F, Guo W, Zhang X, Cao L. Exploring Acute Kidney Injury Incidence in Hip Periprosthetic Joint Infection Treatment With Combined Intravenous and Intra-articular Antibiotic Infusion. Arthroplast Today. 2025 Jan 27;31:101616. doi: 10.1016/j.artd.2025.101616. eCollection 2025 Feb. PMID 39931554
- [Background] Vicenti G, Pesare E, Colasuonno G, Buono C, Albano F, Ladogana T, Passarelli AC, Solarino G. Debridement, Antibiotic Pearls, and Retention of the Implant (DAPRI) in the Treatment of Early Periprosthetic Knee Joint Infections: A Literature Review. Healthcare (Basel). 2024 Apr 16;12(8):843. doi: 10.3390/healthcare12080843. PMID 38667605
- [Background] Perdomo-Lizarraga JC, Combalia A, Fernandez-Valencia JA, Martinez-Pastor JC, Morata L, Soriano A, Munoz-Mahamud E. Long-term implant survival after debridement, antibiotics and implant Retention (DAIR) for acute prosthetic joint infections: is it a viable option beyond four weeks after index arthroplasty? Int Orthop. 2025 Mar;49(3):573-580. doi: 10.1007/s00264-025-06422-6. Epub 2025 Feb 14. PMID 39951052
- [Background] Ayoade F, Li D, Mabrouk A, Todd JR. Periprosthetic Joint Infection. 2023 Oct 14. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK448131/ PMID 28846340
- [Background] Lin S, Villa JM, Rajschmir K, Higuera CA, Grieco P. The Visual Assessment of Cup Position on Anteroposterior Pelvis Radiographs Before Revision Total Hip Arthroplasty for Instability Is Highly Deceiving. Orthopedics. 2025 Jan-Feb;48(1):e22-e26. doi: 10.3928/01477447-20241219-03. Epub 2024 Dec 26. PMID 39724076
- [Background] Li Z. Advancements of biomaterial in hip replacement technology incorporating ceramic materials. J Orthop. 2024 Oct 4;62:27-35. doi: 10.1016/j.jor.2024.09.021. eCollection 2025 Apr. PMID 39473875
- [Background] El Motassime A, Pesare E, Russo A, Salini S, Gava G, Recupero C, Giani T, Covino M, Maccauro G, Vitiello R. The Impact of Frailty and Gender Differences on Hospitalization and Complications in Proximal Femoral Pathological Fractures: A Cross-Sectional Study. J Pers Med. 2024 Sep 18;14(9):991. doi: 10.3390/jpm14090991. PMID 39338245
- [Background] Matrangolo MR, Smimmo A, Vitiello R, De Fazio A, El Motassime A, Noia G, Minutillo F, Maccauro G. Predictor of hip fracture type: a systematic review. Acta Biomed. 2023 Jun 23;94(S2):e2023047. doi: 10.23750/abm.v94iS2.12572. PMID 37366194